CLINICAL TRIAL: NCT05683587
Title: The Effects of Ballet Course on Lower Limb Muscle Strength, Balance and Working Memory of Fitness Studio Students and Their Compliance and Satisfaction With the Course
Brief Title: Effect of Ballet Course on Lower Limb Strength, Balance, Working Memory and the Compliance and Satisfaction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KMUHIRB-E(I)-20220167
Record Dates: First submitted 2022-09-23; First posted 2023-01-13 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2022-09

CONDITIONS: Balance; Lower Limb; Strength; Working Memory; Compliance; Satisfaction
MeSH Terms: conditions — Patient Compliance; Personal Satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): intervention
  Interventions: Other: ballet course, strength course

INTERVENTIONS:
Other: ballet course, strength course — Include of two phase,first phase is strength course for three months and second phase is ballet course for three months.

SUMMARY:
In recent years, sports have become popular, and major gyms or private exercise studios have been opened continuously. A dazzling array of course content allows students to choose according to their preferences. Therefore, how to improve students' compliance with gyms or classrooms, and increase exercise frequency to develop exercise habits , is the current problem faced by the industry.

However, in the case of limited time, the academic side is looking for more effective training courses, and the industry side is trying a variety of courses that are more attractive to the public, hoping to be different from the previous types of sports, improve the motivation of public sports, increase the frequency of exercise and then Maintain exercise habits.

Compared with aerobic dance, boxing, yoga and Pilates, ballet is a niche course, but more and more studies have pointed out that ballet can effectively improve posture, improve lower limb muscle strength, and improve cognitive, executive memory, and working memory.

Therefore, this study intends to explore the effect of ballet courses on lower limb explosiveness, static balance, dynamic balance, cognitive executive function and working memory of exercise studio students. degree and become one of the courses chosen by students for their classes.

ELIGIBILITY:
Inclusion Criteria:

* Studio students willing to participate in the two-stage test.
* Aged between 20 and 64 years old.
* Able to perform test-related movements, including vertical jumping and tiptoe movements.
* No lower extremity musculoskeletal surgery has been performed within six months.

Exclusion Criteria:

* Those who are sick and unable to exercise vigorously under medical advice.
* Those who have studied classical ballet for up to one year.

Ages: 20 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Strength of lower limb | baseline and first month
  Vertical Jump Test
Change from first month Strength of lower limb | first month and second month
  Vertical Jump Test
Change from second month Strength of lower limb | second month and third month
  Vertical Jump Test
Change from third month Strength of lower limb | third month and fourth month
  Vertical Jump Test
Change from fourth month Strength of lower limb | fourth month and fifth month
  Vertical Jump Test
Change from fifth month Strength of lower limb | fifth month and sixth month
  Vertical Jump Test

SECONDARY OUTCOMES:
Change from Baseline static balance | baseline and first month
  Stork Balance Stand Test
Change from first month static balance | first month and second month
  Stork Balance Stand Test
Change from second month static balance | second month and third month
  Stork Balance Stand Test
Change from third month static balance | third month and fourth month
  Stork Balance Stand Test
Change from fourth month static balance | fourth month and fifth month
  Stork Balance Stand Test
Change from fifth month static balance | fifth month and sixth month
  Stork Balance Stand Test
Change from Baseline Dynamic balance | baseline and first month
  Timed-Up-and-Go test
Change from first month Dynamic balance | first month and second month
  Timed-Up-and-Go test
Change from second month Dynamic balance | second month and third month
  Timed-Up-and-Go test
Change from third month Dynamic balance | third month and fourth month
  Timed-Up-and-Go test
Change from fourth month Dynamic balance | fourth month and fifth month
  Timed-Up-and-Go test
Change from fifth month Dynamic balance | fifth month and sixth month
  Timed-Up-and-Go test
Change from Baseline Dynamic balance | baseline and first month
  Y-Balance Test
Change from first month Dynamic balance | first month and second month
  Y-Balance Test
Change from second month Dynamic balance | second month and third month
  Y-Balance Test
Change from third month Dynamic balance | third month and fourth month
  Y-Balance Test
Change from fourth month Dynamic balance | fourth month and fifth month
  Y-Balance Test
Change from fifth month Dynamic balance | fifth month and sixth month
  Y-Balance Test
Change from Baseline Working memory | baseline and third month
  D N-back test
Change from third month Working memory | third month and sixth month
  D N-back test
compliance and satisfaction of ballet and strength courses | sixth month
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lih-Jiun Liaw, Study Chair — Professor
Locations (1):
- Amy Studio fitness studio, Tainan, Taiwan